CLINICAL TRIAL: NCT05790018
Title: Effect of Pregnant Pıllow Used In the Last Trımester on Sleep and Comfort: Randomızed Controlled Study
Brief Title: Effect of Pregnant Pıllow on Sleep and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-betuluzun-001
Record Dates: First submitted 2023-03-01; First posted 2023-03-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy Related; Sleep; Comfort
Keywords: Pregnancy; Pregnancy pillow; Sleep; Comfort

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiment (Experimental): First of all, questionnaire forms and scales will be applied to the pregnant women included in the experimental group in the pre-test (at 29-30 weeks). Then the pregnant pillow will be given and necessary explanations will be given about its use. Second follow-up 33-34. It will be done at the gestational week and the scales will be repeated. The final test is 37-38. It will be done at the gestational week (before birth) and the research will be completed.
  Interventions: Device: PREGNANT PILLOW
- Control (No Intervention): The researcher will apply the questionnaires and scales in the pre-test to the pregnant woman included in the control group, and no other intervention will be applied. 37-38 to the pregnant women in the control group. The final test will be done weekly.

INTERVENTIONS:
Device: PREGNANT PILLOW — First of all, questionnaire forms and scales will be applied to the pregnant women included in the experimental group in the pre-test (at 29-30 weeks). Then the pregnant pillow will be given and necessary explanations will be given about its use. Second follow-up 33-34. It will be done at the gestational week and the scales will be repeated. The final test is 37-38. It will be done at the gestational week (before birth) and the research will be completed.
  Arms: Experiment

SUMMARY:
One of the most special life events of the fertile period is pregnancy. Pregnancy causes many physiological, metabolic, mental and social changes. These changes may adversely affect the sleep quality and comfort levels of pregnant women. Sleep is one of the basic life activities. Comfort is the state of being physiologically, mentally and socially comfortable. The woman who completes her pregnancy comfortably has a high self-confidence and quality of life. On the other hand, it is known that stress, anxiety and depression are experienced more and pregnancy and birth complications increase. For this reason, it is important to determine the comfort levels of pregnant women and to know the factors affecting them. It should not be forgotten that sleep quality in the prenatal period may be effective on the comfort levels of individuals. Evaluation of sleep quality and comfort levels of pregnant women is a routine part of prenatal care. Various interventions can be used to improve the sleep quality of pregnant women. The use of a pregnant pillow in the prenatal period is one of these applications. By providing support and relaxation to 5 different parts of the body simultaneously, the pregnancy pillow helps to increase the sleep quality of expectant mothers during pregnancy and to reduce the neck, abdomen, waist, back and leg pains they experience. It is known that sleep problems are experienced especially in primaries and third trimesters. For this reason, using the pregnant pillow in the third trimester, when sleep problems increase and comfort is adversely affected, may help improve the sleep quality and comfort level of pregnant women. With this planned study, it was aimed to examine the effect of the pregnant pillow used in the last trimester on sleep and comfort.

This research will be carried out with pregnant women who applied to Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital NST and polyclinic unit between 01 March and 31 August 2023. The data of the study will be collected by using Personal Information Form, Information Form on Sleep in Pregnancy, Prenatal Comfort Scale and Pitsburg Sleep Quality Scale.

DETAILED DESCRIPTION:
To research Over 18 years of age Volunteer to participate in the research, Primiparous, 29-30. during pregnancy, Fluent in Turkish, At least primary school graduate, It is planned to include pregnant women who do not have sleep problems, visual/mental and diagnosed psychiatric problems and do not use medication.

Persons who do not meet these criteria and do not volunteer to participate in the study will not be included in the study.

Data Collection The pregnant women included in the study will be randomly assigned to the groups and homogeneity will be ensured in the distribution of the groups. "Random Allocation Software Program" will be used in the randomization of pregnant women into groups and a randomization list for the study will be created. If the pregnant woman leaves the study for any reason during the study, the first pregnant woman who meets the research criteria will be assigned to the other group in the randomization list.

Midwifery Initiative Midwifery Attempts Made to the Control Group The researcher will apply the questionnaires and scales in the pre-test to the pregnant woman included in the control group, and no other intervention will be applied. 37-38 to the pregnant women in the control group. The final test will be done weekly.

Midwifery Attempts Made to the Experimental Group First of all, questionnaire forms and scales will be applied to the pregnant women included in the experimental group in the pre-test (at 29-30 weeks). Then the pregnant pillow will be given and necessary explanations will be given about its use. Second follow-up 33-34. It will be done at the gestational week and the scales will be repeated. The final test is 37-38. It will be done at the gestational week (before birth) and the research will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate the study
* Primiparous
* 29-30. during pregnancy

Exclusion Criteria:

* Sleeping problems
* Vision/mental diagnosed psychiatric problems

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Enrollment: 75 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Prenatal comfort scale | baseline and 4 weeks
  The comfort is one of the primary outcomes. The comfort levels of pregnant women will be measured using the Prenatal Comfort Scale (PCS).
  The PCS consists of 15 items and 5 sub-dimensions. The scale is evaluated over a total of 75 points. It is interpreted that as the score decreases, the comfort level also decreases, and as the score increases, the comfort level also increases.
Pittsburgh sleep quality ındex | baseline and 4 weeks
  Sleep quality is the other primary outcome for this study. Sleep quality of pregnant women will be evaluated with the Pittsburgh Sleep Quality Index (PSQI).
  The PSQI assesses sleep quality and disturbance over the past month. The scale consists of 7 components. Each component is evaluated over 0-3 points. The total score of the 7 components gives the scale total score. The total score ranges from 0 to 21. A total score greater than 5 indicates "poor sleep quality".
Prenatal Comfort Scale (PCS): 2 months | At the end of the 2 months
  From the third trimester, pregnant women will be allowed to sleep on the pregnant pillow. At the end of the 2nd month, PCS will be repeated in order to determine the effect of the pillow used on the sleep and comfort of the pregnant women.
Pittsburgh Sleep Quality Index (PSQI): 2 months | At the end of the 2 months
  From the third trimester, pregnant women will be allowed to sleep on the pregnant pillow. At the end of the 2nd month, PSQI will be repeated in order to determine the effect of the pillow used on the sleep and comfort of the pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya Provincial Health Directorate Sabuncuoğlu Şerefeddin Training and Research Hospital, Amasya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is planned to publish the data obtained from the research in order to enrich the literature.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It will be published after the research is completed.
Access Criteria: Subscribing to the journal in which the article was published